CLINICAL TRIAL: NCT03519542
Title: Muticentric and Prospective Epidemiological Study to Identify Prognosis and Predictive Biomarkers of Response to Angiogenic Drugs Approved in First Line of Treatment for Advanced or Metastatic Renal Cell Carcinoma
Brief Title: Epidemiological Study to Identify Prognosis and Predictive Biomarkers for Advanced or Metastatic Renal Cell Carcinoma
Acronym: SOGANG
Status: Completed | Type: Observational
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Sponsor
Other Study IDs: SOG-ANG-2013-01
Record Dates: First submitted 2014-10-29; First posted 2018-05-09 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib; pazopanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Serum Biomarkers
  * Peripheral Blood
  * Tissue Biomarkers (FFEP tumor tissue from filed tissue sample, protein expresion will be assesed by IHC)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metastatic clear cell renal carcinoma (mRCC) patients: Metastatic clear cell renal carcinoma (mRCC) patients cadidates to receive Sunitinib 50 mg/day 4/2 schedule or Pazopanib 800mg/day until unaccetable toxicity or progression or death under standar clinical practice.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Identify prognosis and predictive biomarkers of response to sunitinib and pazopanib as first line therapy in avanced or metastatic renal cell carcinoma.
  Other Names: Pazopanib

SUMMARY:
Multicentric and prospective epidemiological study (NON INTERVETIONAL) to identify prognosis and predictive biomarkers of response to sunitinib and pazopanib as first line therapy in metstatic renal cell carcinoma.

Molecular determinations will be developed ay CIMA and CNIO.

DETAILED DESCRIPTION:
In coming years new TKIs for the treatment of mRCC are expected to be available. Identificaction of novel biomarkers is required to select those patients who would most benefit from a particular therapeutic strategy:

C-Met is a tyrosine kinase receptor involved in cellular growth and vascular develoment, also identify as a proto-oncogene.

Chemiokines: an increase in pro-angiogenic chemokines such as IL-6 & IL-8 has been also suggested as a tumor dependent possible mechanism influencing invasion and metastasis after anti-VEGF therapy.

PBRM1 (BAF 180) mutation: Second major involved gene in clear cell RCC with truncating mutations in 41% (92/227) of cases. Mutations appear to inactive a protein that plays role in remodeling the structure of genetic material.PBRM1 mutations could be (partially) involved in about 40% of clear cell RCC. PBRM1 may affect the processes of cell divsion in renal cells and could consequently be another target for new drugs.

ELIGIBILITY:
Inclusion Criteria:

* Locally avanced or metastatic renal cell carcinoma with clear-cell component histology candidates to recieve sunitinib or pazopanib in fisrt line under standard clinical practice.
* Measurable disease by CT or MRI
* Life expectancy >3 months
* Written informed consent.
* Performance Status 0-2

Exclusion Criteria:

* Any patients who does not fulfill the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic clear cell renal carcionoma (mCCR) patients candidates to receive sunitinib or pazopanib under standard clinical practice
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Tissue and blood biomarkers | 0 day (pre-treatment), 3month after start of treatment and after progression disease or death or end of study.
  Correlate tissue and blood biomarkers with sunitinib and pazopanib efficacy in terms of progression free survival (PFS) according RECIST criteria.
  Tissue biomarkers: FFEP tumor tissue from filed tissue sample (pre-treatment) Serum biomarkers: 0 day (pre-treatment), 3month after start of treatment and after progression disease or death or end of study.
  Peripheral blood: 0 day (pre-treatment).
Tissue and blood biomarkers | 0 day (pre-treatment), 3month after start of treatment and after progression disease or death or end of study.
  Correlate tissue and blood biomarkers with sunitinib and pazopanib efficacy in terms of overal response rate (ORR) according RECIST criteria.
  Tissue biomarkers: FFEP tumor tissue from filed tissue sample (pre-treatment) Serum biomarkers: 0 day (pre-treatment), 3month after start of treatment and after progression disease or death or end of study.
  Peripheral blood: 0 day (pre-treatment).
Tissue and blood biomarkers | 0 day (pre-treatment), 3month after start of treatment and after progression disease or death or end of study.
  Correlate tissue and blood biomarkers with sunitinib and pazopanib efficacy in terms of overall survival (OS) according RECIST criteria.
  Tissue biomarkers: FFEP tumor tissue from filed tissue sample (pre-treatment) Serum biomarkers: 0 day (pre-treatment), 3month after start of treatment and after progression disease or death or end of study.
  Peripheral blood: 0 day (pre-treatment).
Tumor measure | Under Standar Clinical Practice (every 3 months)
  Tumor measure according RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Esteban, MD. Phd., Principal Investigator — Hospital Universitario Central de Asturias, Spain.
Locations (12):
- Spain (12):
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitarios de Burgos, Burgos
  - Hospital Universiario de León, León
  - Hospital Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico (Madrid), Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Carlos Haya, Málaga
  - Hospital Clínico Lozano Blesa, Zaragoza

REFERENCES:
- See also: Spanish Oncology Genitourinary Group — http://www.sogug.es/